CLINICAL TRIAL: NCT02930876
Title: Feasibility of Home vs. Hospital Based Resistance Training for Advanced Cancer Patients: a Phase II Trial
Brief Title: Feasibility of Home vs. Hospital Based Resistance Training for Advanced Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Calouste Gulbenkian Foundation (Unknown); Centro Hospitalar Lisboa Central (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HR-15/16-2960
Record Dates: First submitted 2016-09-02; First posted 2016-10-12 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2016-08

CONDITIONS: Advanced Cancer
Keywords: sarcopenia; cancer; chemotherapy; palliative care; resistance training
MeSH Terms: conditions — Sarcopenia; Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Resistance training at home (Experimental): Participants will undergo training sessions at their own homes. The exercise program will be individualized and guided by trained physiotherapists, for 3 months completion, aiming at 2-3 sessions a week (27 to 40 sessions in total), each lasting 45-60 minutes.
  Interventions: Behavioral: Resistance training
- Resistance training at the hospital (Experimental): Participants will undergo training sessions at the hospital. The exercise program will be individualized and guided by trained physiotherapists, for 3 months completion, aiming at 2-3 sessions a week (27 to 40 sessions in total), each lasting 45-60 minutes.
  Interventions: Behavioral: Resistance training
- Controls (No Intervention): Participants will be given an information leaflet with the exercise recommendations of the Portuguese national ministry of health.

INTERVENTIONS:
Behavioral: Resistance training — Set of muscle strengthening exercises of all major muscle groups, guided by physiotherapists.
  Arms: Resistance training at home; Resistance training at the hospital

SUMMARY:
Cancer causes 8.2 million deaths each year, with an estimated worldwide cost of $895 billion. Pharmacological treatments provide improvements in expected survival and symptoms, but at cost of a high rate of toxicities and increased time spent by patients away from their homes and families during treatment. This is particularly important for patients with advanced disease as the timeframe at stake relates to their last months of life.

Sarcopenia (i.e. loss of muscle mass together with decreased functional capacity) has been widely reported as an important prognostic factor in advanced cancer, with impact on survival, toxicities, response to treatment and other patient-centered outcomes (such as functional capacity, quality of life and fatigue).

Sarcopenia is a term first used in 1988 by Rosenberg, meaning an age-related loss in skeletal muscle mass and function. It was derived from the greek: sarx = flesh and penia = loss. In 2010, a European Consensus defined sarcopenia as a triad of muscle mass loss, decreased functional performance and muscle strength. It has been reported as a hallmark of cancer, with impact on prognosis, response to treatments, side effects of chemotherapy and recovery after surgery. The prevalence of sarcopenia in advanced cancer seems to vary according to gender, stage, primary tumor location and treatments, being present in about 28 to 67% of patients.

Exercise, in particular resistance training, is one of the most powerful ways of increasing muscle mass and evidence from elderly patients suggests that it is among the most promising interventions for sarcopenia. There is evidence that resistance training can be effective but evidence is still scarce for patients with advanced disease. Historically there have been some concerns regarding safety and efficacy for oncologic patients, and though evidence suggests that resistance training is one of the most preferred forms of exercise by patients, the effectiveness of resistance training alone on sarcopenia in patients with advanced cancer remains unknown. Another question is whether home (which seems to be the patients' preferred location for exercise) produces better results than hospital (the traditional location).

DETAILED DESCRIPTION:
Study hypothesis: Home is the preferred setting for resistance training programs in adults newly diagnosed with advanced cancer, compared to hospital or standard care alone.

AIM: to test the feasibility and clinical impact of home vs. hospital based resistance training programs in adults newly diagnosed with advanced cancer, compared to standard care.

Objective 1: to describe the feasibility (defined as acceptability, compliance, recruitment and retention) of the two intervention models and control; Secondary outcome measures: Objective 2: to test their tolerability (patients' perception) and safety (number of adverse events due to the exercise); Objective 3: to explore the effect of the interventions on clinical outcomes (muscle mass, treatment related toxicities, strength, functional capacity, quality of life, fatigue); Objective 4: to evaluate the associated health resources use (unplanned medical appointments, acute and emergency visits and hospital admissions) in the intervention and control arms.

Study design: the investigators designed a three arm, randomised, open label, phase II trial, in advanced cancer patients, comparing 1) standard treatment concomitant with a resistance training program at home; 2) standard treatment concomitant with a resistance training program at the hospital; 3) standard treatment alone.

Overall trial start date: 01/05/2016 Overall trial end date: 31/03/2017 Condition: Advanced cancer Interventions: Resistance training at home, resistance training at the hospital

ELIGIBILITY:
Inclusion Criteria:

- histological diagnosis of cancer, incurable (stage IIIB/IV according to AJCC 2010).

Exclusion Criteria:

* chemotherapy within 90 days prior to study enrollment
* not having a baseline (pre-treatment) Computed Tomography of the Thorax Abdomen and Pelvis (CTTAP) and whole body dual x-ray absorptometry (DXA) (this is important because having an assessment of baseline muscle mass will allow us to control for baseline sarcopenia and calculate changes from baseline to post-intervention)
* bone metastasis in risk of fracture
* inability to comply with the intervention for any known reasons (including physical or mental impairment that limits the capacity to undertake the exercise program)
* considered to be at cardiovascular risk (defined by a pre-exercise cardiologic evaluation with electrocardiogram (ECG) and echocardiogram when indicated (echocardiogram if >50 years old, NYHA class I, angor, cardiovascular risk factors and abnormal ECG)).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Number of training sessions completed | 3 months after baseline (at the end of the training program)
  Feasibility of the two intervention models assessed by the number of sessions completed
Number of exercises done within each session | 3 months after baseline (at the end of the training program)
  Feasibility of the two intervention models assessed by the number of exercises completed in each session

SECONDARY OUTCOMES:
Tolerability | 3 months after baseline (at the end of the training program)
  Tolerability defined as the patients' perception of whether the program is tolerable on a Likert scale at 3 months after enrollment
Safety of the exercise program | 3 months after baseline (at the end of the training program)
  Evaluated as the number of adverse events due to the exercise program
Change in muscle mass after the 3 months of exercise | Reported at baseline and 3 months after enrolment;
  to explore the effect of the interventions on muscle mass measured by DXA
Frequency of treatment related toxicities | Reported at baseline and 3 months after enrolment;
  to explore the effect of the interventions on treatment related toxicities reported according to Common Toxicity Criteria for Adverse Events
Change in strength after the 3 months of exercise | Reported at baseline and 3 months after enrolment;
  to explore the effect of the interventions on strength assessed through sit to stand transitions
Change in functional capacity after the 3 months of exercise vs controls | Reported at baseline and 3 months after enrolment;
  to explore the effect of the interventions on functional capacity assessed though 6 minute walking test
Change in quality of life after the 3 months of exercise vs controls | Reported at baseline and 3 months after enrolment;
  to explore the effect of the interventions on quality of life assessed using EORTC QoL C30
Change in fatigue after the 3 months of fatigue vs controls | Reported at baseline and 3 months after enrolment;
  to explore the effect of the interventions on fatigue assessed using Brief Fatigue Inventory
Health resources use | 3 months after baseline (at the end of the training program)
  number of unplanned medical appointments, acute and emergency visits and hospital admissions

CONTACTS AND LOCATIONS:
Locations (1):
- King's College of London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Presentation in conferences and publication in peer reviewed journals

REFERENCES:
- [Derived] Ribeiro C, Santos R, Correia P, Maddocks M, Gomes B. Resistance training in advanced cancer: a phase II safety and feasibility trial-home versus hospital. BMJ Support Palliat Care. 2022 Sep;12(3):287-291. doi: 10.1136/bmjspcare-2020-002230. Epub 2020 Aug 13. PMID 32792420